CLINICAL TRIAL: NCT04826900
Title: A Randomized Control Trial to Compare the Effects Between Wearable Robotic System and Robotic Mirror Therapy in Patients With Spastic Hemiplegia Post Botulinum Toxin Injection: Neurophysiological and Behavior Outcomes
Brief Title: Wearable Robotic System and Robotic Mirror Therapy in Spastic Hemiplegia Post Botulinum Toxin Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRMPG8J0211
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2021-03

CONDITIONS: Hemiplegia, Spastic; Spastic
Keywords: Stroke rehabilitation; Spasticity; Botulinum toxin type A injection; Mirror therapy; Robot
MeSH Terms: conditions — Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant
Masking Description: There will be a research code representing patients' identity, this code will not show patients' name, social security number, and home address. For the results of patients' visit and the diagnosis, the study moderator will maintain a confidential attitude and be careful to maintain patients' privacy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Group (Experimental): Training session included 45 minutes Robotic Therapy, followed by 15-minute functional training. The robotic group will receive 3 sessions per week, for 8 weeks.
  Interventions: Procedure: BoNT-A injections; Other: Robotic therapy (RT); Other: Functional task training
- Robotic Mirror Group (Experimental): Training session included 45 minutes Robotic Mirror Therapy, followed by 15-minute functional training. The robotic group will receive 3 sessions per week, for 8 weeks.
  Interventions: Procedure: BoNT-A injections; Other: Robotic mirror therapy (RMT); Other: Functional task training

INTERVENTIONS:
Procedure: BoNT-A injections — Botox brand BoNT-A Purified Neurotoxin Complex, (Allergan Pharmaceuticals, Irvine, CA) will be prepared by diluting lyophilized toxin with 0.9% saline to a concentration of 33-100 U/ml. depending on the size of the target muscle. Location of the targeted muscle will be confirmed by using echo guide. The total dose range is 200 units to 500 units. The dose range of each target muscle is as below: 20 and 75 units for flexor carpi ulnaris and flexor carpi radials; 12.5-35 units per fascicle in the flexor digitorum sublimis and flexor digitorum profundus (maximum dose: 120 units for each of these muscles); 10-35 units in the flexor pollicis longus; 25-100 units in the brachioradial ; 50-200 units in the biceps brachii; and 25-75 units in the pronator teres
Other: Robotic therapy (RT) — A wearable robotic hand system will be used in this study. The robotic hand system consisted with a wearable exoskeletal hand, sensor glove, and a control box. On the exoskeletal hand, there are five actuators on each of finger structure that can provide external power to bring individual finger moving. The sensor glove has five sensors that can detect the finger's posture during movement and then manipulates exoskeletal hand via the control box. The patient's unaffected hand wears the sensor glove, the affected hand wears the wearable exoskeleton hand, and the unaffected hand does the certain transitive and intransitive tasks as the mirror group, and then makes the affected hand do the same movements driven by the exoskeleton robotic hand.
  Arms: Robotic Group
Other: Robotic mirror therapy (RMT) — Wearable robotic hand system and mirror system will be used in this group.. The patients in the group will wear the robotic hand to do the mirror therapy. The patient's unaffected hand wears the sensor glove, the affected hand wears the wearable exoskeletal hand, a mirror box with a mirror will be placed in the patient 's midsagittal plane beside the unaffected hand to block his or her view of the affected hand. The patient's unaffected hand does the certain transitive and intransitive tasks and the patient will be instructed to look at the reflection of the unaffected hand in the mirror as if it is the affected hand (the visual input). At the same time the affected hand will be passively moved by the exoskeleton robotic hand which is under the .control of the unaffected hand.
  Arms: Robotic Mirror Group
Other: Functional task training — After either 45 minutes of RT or RMT, all participants receive 15 minutes of training in functional tasks. The functional tasks included taking up and holding bowl or using eating utensils , bringing a cup for drinking, drying sucks by clips, open ing or closing door , turning on or off the light, cleaning the table or window and so on . The functional tasks training will be bases on the needs and ability of patients.

SUMMARY:
The purpose of this project is to examine and compare the immediate and long-term effects of combined Botulinum toxin type A(BoNT-A) injection with wearable robotic hand system (RT) and Robotic mirror therapy (RMT) in patients with spastic hemiplegic stroke.

DETAILED DESCRIPTION:
Spasticity, a common impairment after stroke, has a profound impact on activity and participation for patients. BoNT-A injection combined with rehabilitation training is recommended to enhance functional recovery of patients with spastic hemiplegic stroke.

Patients with spasticity usually have lower motor function and worse sensory deficits than patients without spasticity. Designing the post BoNT-A injection rehabilitation program should consider the above issues. RT and MT are two interventions providing sensorimotor input for patient with low motor function. Combining both approaches (wearing robotic hand to do mirror therapy) might facilitate the sensorimotor cortex that controls movement and might augment somatosensory input and further treatment efficacy. It is unknown whether and how combining BoNT injection with bilateral RT vs with MT vs with RMT engenders differential effects on motor and related functional performance in patients with spastic hemiplegic stroke.

Forty-eight participants with chronic spastic hemiplegic stroke will be recruited and randomly assigned to one of 2 groups: RT, and RMT. All the post- injection interventions will be implemented 60 minutes/day, 3 days/week, for 8 weeks. At each training session all patients will receive 45-minute RT, or RMT, then 15-minute functional task training.

The outcome measures include 1) body function and structures: Fugl-Meyer Assessment, Modified Ashworth Scale, Medical Research Council scale, 2) activity and participation: Box and block test, Motor Activity Log, and Nottingham Extended Activities of Daily Living Scale, Action Research Arm Test. In addition, to directly reflect a patient's unique needs and goals, Goal Attainment Scaling will be assessed. Electroencephalography (EEG) and functional near infrared reflectance spectroscopy (NIRS) assessments will be done to assess the neurophysiologic effects of the 3 kinds of intervention. The outcome will be measured at pre-treatment,1-week after BoNT-A injection, post-treatment, and 3-month follow- up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and imagine diagnosis of a first or recurrent unilateral stroke ≥ 3 months
* Finger flexor muscles spasticity (modified Ashworth scale of ≥ 1+)
* Initial motor part of UE of FMA score ranging from 10 to 56 indicating moderate to severe movement impairment
* No serious cognitive impairment (i.e., Mini Mental State Exam score > 20)
* Age ≥ 20 years

Exclusion Criteria:

* Pregnant
* With bilateral hemispheric or cerebellar lesions
* Sever aphasia
* Significant visual field deficits or hemineglect
* Contraindication for BoNT-A injection
* Treatment with BoNT-A within 6 months before recruitment
* Any fixed joint contracture of the affected upper limb
* A history of orthopedic or other neurological diseases and/or medical conditions that would prevent adherence to the rehabilitation protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-01-23 (Actual); Study Completion 2022-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hung Jen-Wen, Principal Investigator — Chang Gung Memorial Hospital-Kaohsiung Medical Center
Locations (1):
- Department of Rehabilitation, Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ada L, O'Dwyer N, O'Neill E. Relation between spasticity, weakness and contracture of the elbow flexors and upper limb activity after stroke: an observational study. Disabil Rehabil. 2006 Jul 15-30;28(13-14):891-7. doi: 10.1080/09638280500535165. PMID 16777777
- [Background] Amano S, Takebayashi T, Hanada K, Umeji A, Marumoto K, Furukawa K, Domen K. Constraint-Induced Movement Therapy After Injection of Botulinum Toxin Type A for a Patient With Chronic Stroke: One-Year Follow-up Case Report. Phys Ther. 2015 Jul;95(7):1039-45. doi: 10.2522/ptj.20140329. Epub 2015 Jan 15. PMID 25592185
- [Background] Bhakta BB, Cozens JA, Chamberlain MA, Bamford JM. Impact of botulinum toxin type A on disability and carer burden due to arm spasticity after stroke: a randomised double blind placebo controlled trial. J Neurol Neurosurg Psychiatry. 2000 Aug;69(2):217-21. doi: 10.1136/jnnp.69.2.217. PMID 10896696
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Brewer BR, McDowell SK, Worthen-Chaudhari LC. Poststroke upper extremity rehabilitation: a review of robotic systems and clinical results. Top Stroke Rehabil. 2007 Nov-Dec;14(6):22-44. doi: 10.1310/tsr1406-22. PMID 18174114
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Carswell A, McColl MA, Baptiste S, Law M, Polatajko H, Pollock N. The Canadian Occupational Performance Measure: a research and clinical literature review. Can J Occup Ther. 2004 Oct;71(4):210-22. doi: 10.1177/000841740407100406. PMID 15586853
- [Background] Chuang LL, Wu CY, Lin KC. Reliability, validity, and responsiveness of myotonometric measurement of muscle tone, elasticity, and stiffness in patients with stroke. Arch Phys Med Rehabil. 2012 Mar;93(3):532-40. doi: 10.1016/j.apmr.2011.09.014. Epub 2012 Jan 4. PMID 22222143
- [Background] de Paiva A, Meunier FA, Molgo J, Aoki KR, Dolly JO. Functional repair of motor endplates after botulinum neurotoxin type A poisoning: biphasic switch of synaptic activity between nerve sprouts and their parent terminals. Proc Natl Acad Sci U S A. 1999 Mar 16;96(6):3200-5. doi: 10.1073/pnas.96.6.3200. PMID 10077661
- [Background] Dedding C, Cardol M, Eyssen IC, Dekker J, Beelen A. Validity of the Canadian Occupational Performance Measure: a client-centred outcome measurement. Clin Rehabil. 2004 Sep;18(6):660-7. doi: 10.1191/0269215504cr746oa. PMID 15473118
- [Background] Demetrios M, Khan F, Turner-Stokes L, Brand C, McSweeney S. Multidisciplinary rehabilitation following botulinum toxin and other focal intramuscular treatment for post-stroke spasticity. Cochrane Database Syst Rev. 2013 Jun 5;2013(6):CD009689. doi: 10.1002/14651858.CD009689.pub2. PMID 23740539
- [Background] Elia AE, Filippini G, Calandrella D, Albanese A. Botulinum neurotoxins for post-stroke spasticity in adults: a systematic review. Mov Disord. 2009 Apr 30;24(6):801-12. doi: 10.1002/mds.22452. PMID 19224614
- [Background] Esquenazi A, Novak I, Sheean G, Singer BJ, Ward AB. International consensus statement for the use of botulinum toxin treatment in adults and children with neurological impairments--introduction. Eur J Neurol. 2010 Aug;17 Suppl 2:1-8. doi: 10.1111/j.1468-1331.2010.03125.x. PMID 20633176
- [Background] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Background] Foley N, Pereira S, Salter K, Fernandez MM, Speechley M, Sequeira K, Miller T, Teasell R. Treatment with botulinum toxin improves upper-extremity function post stroke: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2013 May;94(5):977-89. doi: 10.1016/j.apmr.2012.12.006. Epub 2012 Dec 19. PMID 23262381
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Gompertz, P., Pound, P., Ebrahim, S. (1994). Validity of the extended activities of daily living scale. Clinical Rehabilitation, 8, 275-280.
- [Background] Gordon JE, Powell C, Rockwood K. Goal attainment scaling as a measure of clinically important change in nursing-home patients. Age Ageing. 1999 May;28(3):275-81. doi: 10.1093/ageing/28.3.275. PMID 10475864
- [Background] Gregson JM, Leathley MJ, Moore AP, Smith TL, Sharma AK, Watkins CL. Reliability of measurements of muscle tone and muscle power in stroke patients. Age Ageing. 2000 May;29(3):223-8. doi: 10.1093/ageing/29.3.223. PMID 10855904
- [Background] Hsieh YW, Wu CY, Liao WW, Lin KC, Wu KY, Lee CY. Effects of treatment intensity in upper limb robot-assisted therapy for chronic stroke: a pilot randomized controlled trial. Neurorehabil Neural Repair. 2011 Jul-Aug;25(6):503-11. doi: 10.1177/1545968310394871. Epub 2011 Mar 24. PMID 21436390
- [Background] Krebs HI, Volpe BT, Williams D, Celestino J, Charles SK, Lynch D, Hogan N. Robot-aided neurorehabilitation: a robot for wrist rehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2007 Sep;15(3):327-35. doi: 10.1109/TNSRE.2007.903899. PMID 17894265
- [Background] Kwakkel G, Kollen BJ, Krebs HI. Effects of robot-assisted therapy on upper limb recovery after stroke: a systematic review. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):111-21. doi: 10.1177/1545968307305457. Epub 2007 Sep 17. PMID 17876068
- [Background] Lance JW. The control of muscle tone, reflexes, and movement: Robert Wartenberg Lecture. Neurology. 1980 Dec;30(12):1303-13. doi: 10.1212/wnl.30.12.1303. No abstract available. PMID 7192811
- [Background] Levy CE, Giuffrida C, Richards L, Wu S, Davis S, Nadeau SE. Botulinum toxin a, evidence-based exercise therapy, and constraint-induced movement therapy for upper-limb hemiparesis attributable to stroke: a preliminary study. Am J Phys Med Rehabil. 2007 Sep;86(9):696-706. doi: 10.1097/PHM.0b013e31813e2b4d. PMID 17709993
- [Background] Bayley M, Lindsay P, Hellings C, Woodbury E, Phillips S; Canadian Stroke Strategy (a joint initiative of the Canadian Stroke Network and the Heart and Stroke Foundation of Canada). Balancing evidence and opinion in stroke care: the 2008 best practice recommendations. CMAJ. 2008 Dec 2;179(12):1247-9. doi: 10.1503/cmaj.081536. No abstract available. PMID 19047599
- [Background] Luft AR, McCombe-Waller S, Whitall J, Forrester LW, Macko R, Sorkin JD, Schulz JB, Goldberg AP, Hanley DF. Repetitive bilateral arm training and motor cortex activation in chronic stroke: a randomized controlled trial. JAMA. 2004 Oct 20;292(15):1853-61. doi: 10.1001/jama.292.15.1853. PMID 15494583
- [Background] Medical Research Council. (1976). Aids to examination of the peripheral nervous system. Memorandum no. 45. London: Her Majesty's Stationary Office.
- [Background] Michielsen ME, Selles RW, van der Geest JN, Eckhardt M, Yavuzer G, Stam HJ, Smits M, Ribbers GM, Bussmann JB. Motor recovery and cortical reorganization after mirror therapy in chronic stroke patients: a phase II randomized controlled trial. Neurorehabil Neural Repair. 2011 Mar-Apr;25(3):223-33. doi: 10.1177/1545968310385127. Epub 2010 Nov 4. PMID 21051765
- [Background] Michielsen ME, Smits M, Ribbers GM, Stam HJ, van der Geest JN, Bussmann JB, Selles RW. The neuronal correlates of mirror therapy: an fMRI study on mirror induced visual illusions in patients with stroke. J Neurol Neurosurg Psychiatry. 2011 Apr;82(4):393-8. doi: 10.1136/jnnp.2009.194134. Epub 2010 Sep 22. PMID 20861065
- [Background] Morris DM, Uswatte G, Crago JE, Cook EW 3rd, Taub E. The reliability of the wolf motor function test for assessing upper extremity function after stroke. Arch Phys Med Rehabil. 2001 Jun;82(6):750-5. doi: 10.1053/apmr.2001.23183. PMID 11387578
- [Background] Nouri, F.M., Lincoln, N.B. (1987). An extended activities of daily living scale for stroke patients. Clinical Rehabilitation, 1, 301-305.
- [Background] Pandyan AD, Johnson GR, Price CI, Curless RH, Barnes MP, Rodgers H. A review of the properties and limitations of the Ashworth and modified Ashworth Scales as measures of spasticity. Clin Rehabil. 1999 Oct;13(5):373-83. doi: 10.1191/026921599677595404. PMID 10498344
- [Background] Park SW, Wolf SL, Blanton S, Winstein C, Nichols-Larsen DS. The EXCITE Trial: Predicting a clinically meaningful motor activity log outcome. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):486-93. doi: 10.1177/1545968308316906. PMID 18780883
- [Background] Pennati GV, Da Re C, Messineo I, Bonaiuti D. How could robotic training and botolinum toxin be combined in chronic post stroke upper limb spasticity? A pilot study. Eur J Phys Rehabil Med. 2015 Aug;51(4):381-7. Epub 2014 Oct 31. PMID 25358636
- [Background] Platz T, Pinkowski C, van Wijck F, Kim IH, di Bella P, Johnson G. Reliability and validity of arm function assessment with standardized guidelines for the Fugl-Meyer Test, Action Research Arm Test and Box and Block Test: a multicentre study. Clin Rehabil. 2005 Jun;19(4):404-11. doi: 10.1191/0269215505cr832oa. PMID 15929509
- [Background] Portney, L. G., & Watkins, M. P. (2009). Power and sample size. Foundations of clinical research: Applications to practice (3rd ed., pp. 705-719). Upper Saddle River, N.J.: Pearson/Prentice Hall.
- [Background] Prange GB, Jannink MJ, Groothuis-Oudshoorn CG, Hermens HJ, Ijzerman MJ. Systematic review of the effect of robot-aided therapy on recovery of the hemiparetic arm after stroke. J Rehabil Res Dev. 2006 Mar-Apr;43(2):171-84. doi: 10.1682/jrrd.2005.04.0076. PMID 16847784
- [Background] Rockwood K, Stolee P, Fox RA. Use of goal attainment scaling in measuring clinically important change in the frail elderly. J Clin Epidemiol. 1993 Oct;46(10):1113-8. doi: 10.1016/0895-4356(93)90110-m. PMID 8410096
- [Background] Schasfoort FC, Bussmann JB, Martens WL, Stam HJ. Objective measurement of upper limb activity and mobility during everyday behavior using ambulatory accelerometry: the upper limb activity monitor. Behav Res Methods. 2006 Aug;38(3):439-46. doi: 10.3758/bf03192798. PMID 17186754
- [Background] Sheean GL. Botulinum treatment of spasticity: why is it so difficult to show a functional benefit? Curr Opin Neurol. 2001 Dec;14(6):771-6. doi: 10.1097/00019052-200112000-00015. PMID 11723387
- [Background] Sheean G, Lannin NA, Turner-Stokes L, Rawicki B, Snow BJ; Cerebral Palsy Institute. Botulinum toxin assessment, intervention and after-care for upper limb hypertonicity in adults: international consensus statement. Eur J Neurol. 2010 Aug;17 Suppl 2:74-93. doi: 10.1111/j.1468-1331.2010.03129.x. PMID 20633180
- [Background] Stevens JA, Stoykov ME. Using motor imagery in the rehabilitation of hemiparesis. Arch Phys Med Rehabil. 2003 Jul;84(7):1090-2. doi: 10.1016/s0003-9993(03)00042-x. PMID 12881842
- [Background] Stinear CM, Barber PA, Coxon JP, Fleming MK, Byblow WD. Priming the motor system enhances the effects of upper limb therapy in chronic stroke. Brain. 2008 May;131(Pt 5):1381-90. doi: 10.1093/brain/awn051. Epub 2008 Mar 20. PMID 18356189
- [Background] Stoykov ME, Stinear JW. Active-passive bilateral therapy as a priming mechanism for individuals in the subacute phase of post-stroke recovery: a feasibility study. Am J Phys Med Rehabil. 2010 Nov;89(11):873-8. doi: 10.1097/PHM.0b013e3181f1c31c. PMID 20736818
- [Background] Sun SF, Hsu CW, Sun HP, Hwang CW, Yang CL, Wang JL. Combined botulinum toxin type A with modified constraint-induced movement therapy for chronic stroke patients with upper extremity spasticity: a randomized controlled study. Neurorehabil Neural Repair. 2010 Jan;24(1):34-41. doi: 10.1177/1545968309341060. Epub 2009 Sep 3. PMID 19729582
- [Background] Takekawa T, Abo M, Ebihara K, Taguchi K, Sase Y, Kakuda W. Long-term effects of injection of botulinum toxin type A combined with home-based functional training for post-stroke patients with spastic upper limb hemiparesis. Acta Neurol Belg. 2013 Dec;113(4):469-75. doi: 10.1007/s13760-013-0208-4. Epub 2013 May 29. PMID 23716062
- [Background] Taub, E., Crago, J., & Uswatte, G. (1998). Constraint-induced movement therapy: A new approach to teatment in physical medicine. Rehabilitation Psychology, 43, 152-170.
- [Background] Teng EL, Chui HC. The Modified Mini-Mental State (3MS) examination. J Clin Psychiatry. 1987 Aug;48(8):314-8. PMID 3611032
- [Background] European Stroke Organisation (ESO) Executive Committee; ESO Writing Committee. Guidelines for management of ischaemic stroke and transient ischaemic attack 2008. Cerebrovasc Dis. 2008;25(5):457-507. doi: 10.1159/000131083. Epub 2008 May 6. PMID 18477843
- [Background] Thielman G, Kaminski T, Gentile AM. Rehabilitation of reaching after stroke: comparing 2 training protocols utilizing trunk restraint. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):697-705. doi: 10.1177/1545968308315998. PMID 18971384
- [Background] Turner-Stokes L. Goal attainment scaling (GAS) in rehabilitation: a practical guide. Clin Rehabil. 2009 Apr;23(4):362-70. doi: 10.1177/0269215508101742. Epub 2009 Jan 29. PMID 19179355
- [Background] Urbaniak, G. C., & Plous, S. (2013). Research Randomizer (Version 4.0) [Computer software]. Retrieved June 22, 2013, from http://www.randomizer.org/
- [Background] Uswatte G, Foo WL, Olmstead H, Lopez K, Holand A, Simms LB. Ambulatory monitoring of arm movement using accelerometry: an objective measure of upper-extremity rehabilitation in persons with chronic stroke. Arch Phys Med Rehabil. 2005 Jul;86(7):1498-501. doi: 10.1016/j.apmr.2005.01.010. PMID 16003690
- [Background] Uswatte G, Giuliani C, Winstein C, Zeringue A, Hobbs L, Wolf SL. Validity of accelerometry for monitoring real-world arm activity in patients with subacute stroke: evidence from the extremity constraint-induced therapy evaluation trial. Arch Phys Med Rehabil. 2006 Oct;87(10):1340-5. doi: 10.1016/j.apmr.2006.06.006. PMID 17023243
- [Background] Uswatte, G., Taub, E. Constraint-induced movement therapy: new approaches to outcome measurement in rehabilitation. In: Stuss DT, Winocur G, Robertson IH, editors. Cognitive neurorehabilitation: A comprehensive approach. Cambridge: Cambridge Univ Pr; 1999. p 215-29.
- [Background] Uswatte G, Taub E, Morris D, Light K, Thompson PA. The Motor Activity Log-28: assessing daily use of the hemiparetic arm after stroke. Neurology. 2006 Oct 10;67(7):1189-94. doi: 10.1212/01.wnl.0000238164.90657.c2. PMID 17030751
- [Background] Vain, A. (1995). Estimation of the functional state of skeletal muscle. In P. H. Veltink & H. B. K. Boom (Eds.), Control of ambulation using functional neuromuscular stimulation (pp. 51-55). Enschede: University of Twente Press.
- [Background] van der Lee JH, Beckerman H, Knol DL, de Vet HC, Bouter LM. Clinimetric properties of the motor activity log for the assessment of arm use in hemiparetic patients. Stroke. 2004 Jun;35(6):1410-4. doi: 10.1161/01.STR.0000126900.24964.7e. Epub 2004 Apr 15. PMID 15087552
- [Background] Watkins CL, Leathley MJ, Gregson JM, Moore AP, Smith TL, Sharma AK. Prevalence of spasticity post stroke. Clin Rehabil. 2002 Aug;16(5):515-22. doi: 10.1191/0269215502cr512oa. PMID 12194622
- [Background] Welmer AK, von Arbin M, Widen Holmqvist L, Sommerfeld DK. Spasticity and its association with functioning and health-related quality of life 18 months after stroke. Cerebrovasc Dis. 2006;21(4):247-53. doi: 10.1159/000091222. Epub 2006 Jan 27. PMID 16446538
- [Background] Whitall J, Savin DN Jr, Harris-Love M, Waller SM. Psychometric properties of a modified Wolf Motor Function test for people with mild and moderate upper-extremity hemiparesis. Arch Phys Med Rehabil. 2006 May;87(5):656-60. doi: 10.1016/j.apmr.2006.02.004. PMID 16635628
- [Background] Wissel J, Schelosky LD, Scott J, Christe W, Faiss JH, Mueller J. Early development of spasticity following stroke: a prospective, observational trial. J Neurol. 2010 Jul;257(7):1067-72. doi: 10.1007/s00415-010-5463-1. Epub 2010 Feb 6. PMID 20140444
- [Background] Wu CY, Chuang LL, Lin KC, Horng YS. Responsiveness and validity of two outcome measures of instrumental activities of daily living in stroke survivors receiving rehabilitative therapies. Clin Rehabil. 2011 Feb;25(2):175-83. doi: 10.1177/0269215510385482. Epub 2010 Nov 8. PMID 21059664
- [Background] Wu CY, Huang PC, Chen YT, Lin KC, Yang HW. Effects of mirror therapy on motor and sensory recovery in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2013 Jun;94(6):1023-30. doi: 10.1016/j.apmr.2013.02.007. Epub 2013 Feb 15. PMID 23419791
- [Background] Yen JT, Li S. Altered force perception in stroke survivors with spastic hemiplegia. J Rehabil Med. 2015 Nov;47(10):917-23. doi: 10.2340/16501977-2019. PMID 26550912
- [Derived] Hung JW, Chen YJ, Wu WC, Chou CX, Chang HF, Yu MY, Chen PC, Guo TM. Botulinum toxin A combining with robot-assisted bimanual therapy integrating mirror therapy versus botulinum toxin A combining with robot-assisted bimanual therapy in patients with post-stroke spastic fingers: a randomized controlled pilot trial. J Neuroeng Rehabil. 2025 Oct 28;22(1):224. doi: 10.1186/s12984-025-01761-2. PMID 41152923

RESULTS

PARTICIPANT FLOW:
Groups:
- Robotic Group: Training session included 45 minutes Robotic Therapy, followed by 15-minute functional training. The robotic group will receive 3 sessions per week, for 8 weeks.
  BoNT-A injections: Botox brand BoNT-A Purified Neurotoxin Complex, will be prepared by diluting lyophilized toxin with 0.9% saline to a concentration of 33-100 U/ml. depending on the size of the target muscle. Location of the targeted muscle will be confirmed by using echo guide. The total dose range is 200 units to 500 units. The dose range of each target muscle is as below: 20 and 75 units for flexor carpi ulnaris and flexor carpi radials; 12.5-35 units per fascicle in the flexor digitorum sublimis and flexor digitorum profundus (maximum dose: 120 units for each of these muscles); 10-35 units in the flexor pollicis longus; 25-100 units in the brachioradial ; 50-200 units in the biceps brachii; and 25-75 units in the pronator teres
  Robotic therapy (RT): A wearable robotic hand system will be used in this study. The robotic hand system consisted with a wearable exoskeletal hand, sensor glove, and a control box.
  Functional task training: After either 45 minutes of RT or RMT, all participants receive 15 minutes of training in functional tasks. The functional tasks training will be bases on the needs and ability of patients.
- Robotic Mirror Group: Training session included 45 minutes Robotic Mirror Therapy, followed by 15-minute functional training. The robotic group will receive 3 sessions per week, for 8 weeks.
  BoNT-A injections: Botox brand BoNT-A Purified Neurotoxin Complex, (Allergan Pharmaceuticals, Irvine, CA) will be prepared by diluting lyophilized toxin with 0.9% saline to a concentration of 33-100 U/ml. depending on the size of the target muscle. Location of the targeted muscle will be confirmed by using echo guide. The total dose range is 200 units to 500 units. The dose range of each target muscle is as below: 20 and 75 units for flexor carpi ulnaris and flexor carpi radials; 12.5-35 units per fascicle in the flexor digitorum sublimis and flexor digitorum profundus (maximum dose: 120 units for each of these muscles); 10-35 units in the flexor pollicis longus; 25-100 units in the brachioradial ; 50-200 units in the biceps brachii; and 25-75 units in the pronator teres
  Robotic mirror therapy (RMT): Wearable robotic hand system and mirror system will be used in this group.The patients in the group will wear the robotic hand to do the mirror therapy.
  Functional task training: After either 45 minutes of RMT, all participants receive 15 minutes of training in functional tasks.The functional tasks training will be bases on the needs and ability of patients.
Period: Overall Study
Arm/Group | Robotic Group | Robotic Mirror Group
Started | 15 | 16
Completed | 14 | 15
Not Completed | 1 | 1
Not completed — Family factor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robotic Group | Robotic Mirror Group | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.07 (10.36) | 48.60 (9.65) | 47.86 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  Taiwan | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment (FMA)
Description: Fugl-Meyer Assessment for Upper Extremity (FMA-UE): The FMA-UE was used to assess the patient's reflexes, movements, and coordination of upper limbs. It consists of 33 items scored on a 3-point ordinal scale (0, cannot perform; 1, performs partially; 2, performs fully). (Fugl-Meyer, Jääskö, Leyman, Olsson, & Steglind, 1975) . The total score ranges from 0 to 66, and a higher score indicates better motor function. Satisfactory psychometric properties of the FMA have been demonstrated. (Thomas Platz et al., 2005).
Time Frame: Change from baseline at 5 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic Group | Robotic Mirror Group
Number analyzed (Participants) | 14 | 15
score on a scale | 3 [-0.25 to 8.25] | 6 [5 to 9]

2. Primary Outcome: Medical Research Council Scale (MRC)
Description: The MRC scale will be used to examine the muscle strength of the affected arm (Medical Research Council, 1976). The MRC scale is a reliable measurement which ranges from 0 (no contraction) to 5 (normal power). The muscle strength will be measured at the shoulder flexor/abductor, elbow flexors/extensors, wrist flexors/extensors, and finger flexors/extensors by using the MRC in this project. Total scale combines all range and computes average scores. Flexor scale combines elbow flexors, wrist flexors, fingers flexors and computes average scores. Proximal scale combines shoulder flexor/abductor, elbow flexors/extensors, and computes average scores. Distal scale combines wrist flexors/extensors, and finger flexors/extensors. The higher scores mean a better outcome.
Time Frame: Change from baseline at 5 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic Group | Robotic Mirror Group
Number analyzed (Participants) | 14 | 15
score on a scale
  Total | 0.30 [0.03 to 0.71] | 0.35 [0.20 to 0.60]
  Flexor | 0.17 [-0.17 to 0.50] | 0.17 [0.00 to 0.50]
  Finger Flexor | 0.25 [0.00 to 0.50] | 0.50 [0.00 to 1.00]
  Finger Extensor | 0.25 [0.00 to 0.63] | 0.00 [0.00 to 1.00]
  Proximal | 0.33 [-0.19 to 0.60] | 0.42 [0.25 to 0.50]
  Distal | 0.40 [0.00 to 0.75] | 0.42 [0.13 to 0.63]

3. Primary Outcome: Modified Ashworth Scale (MAS)
Description: Spasticity of skeletal muscle in upper extremity was evaluated by using the MAS scale. It uses a 8-point scale(0, 1, 1.5, 2, 2.5, 3, 3.5, 4) to score the average resistance to passive movement for each join with higher score indicating higher spasticity. The MAS has shown good reliability and validity. We assessed the MAS of shoulder flexor/extensor/abductor/adductor, elbow flexors/extensors, forearm pronator/supinator, wrist flexors/extensors, and finger flexors/extensors in this project. Total scale combines all range and computes average scores. Flexor scale combines elbow extensor, wrist extensor, fingers extensor and computes average scores. Proximal scale combines shoulder flexor/extensor/abductor/adductor, elbow flexors/extensors and computes average scores. Distal scale combines forearm pronator/supinator, wrist flexors/extensors, and finger flexors/extensors. The maximum of MAS scale is 4, and the minimum is 0. The higher scores mean a worse outcome.
Time Frame: Change from baseline at 5 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic Group | Robotic Mirror Group
Number analyzed (Participants) | 14 | 15
score on a scale
  Total | -0.33 [-0.36 to -0.16] | -0.17 [-0.25 to -0.08]
  Flexor | -0.42 [-0.67 to 0.00] | -0.17 [-0.33 to 0.00]
  Finger Flexor | -0.25 [-0.63 to 0.50] | 0.00 [-0.50 to 0.00]
  Proximal | -0.17 [-0.29 to -0.06] | -0.08 [-0.25 to -0.08]
  Distal | -0.38 [-0.69 to -0.15] | -0.33 [-0.42 to -0.25]

4. Primary Outcome: Box and Block Test (BBT)
Description: The BBT, which evaluates manual dexterity of the paretic UE, uses a wooden box that has two equally sized compartments. Cubes were placed in one compartment, and the participants were instructed to move the cubes to the other compartment one by one and as quickly as possible within 60 seconds. The score was determined by calculating the number of cubes carried across the partition. The BBT has high test-retest reliability in participants with stroke(Thomas Platz et al., 2005).
Time Frame: Change from baseline at 5 months
Measure: Median (Inter-Quartile Range); unit: cubes/minute
Arm/Group | Robotic Group | Robotic Mirror Group
Number analyzed (Participants) | 14 | 15
cubes/minute | 0 [0 to 1.25] | 0 [0 to 1]

5. Primary Outcome: Motor Activity Log (MAL) - Amount of Use Scale (AOU)
Description: The MAL is a semi-structured interview to rate how much [amount of use scale (AOU)] they use their affected upper extremity in 30 daily activities using a 6-point scale. Higher scores represent better performance. The MAL has established reliability, validity, and responsiveness in patients with stroke. The MAL will be used to measure daily use of the affected upper limb in daily life in this project.The total score ranges from 0 to 30.
Time Frame: Change from baseline at 5 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic Group | Robotic Mirror Group
Number analyzed (Participants) | 14 | 15
score on a scale | 0.14 [-0.02 to 0.64] | 0.34 [0.05 to 0.96]

6. Primary Outcome: Motor Activity Log (MAL) - Quality of Movement Scale (QOM)
Description: The MAL is a semi-structured interview to rate how well [quality of movement scale (QOM)] they use their affected upper extremity in 30 daily activities using a 6-point scale. Higher scores represent better performance. The MAL has established reliability, validity, and responsiveness in patients with stroke. The MAL will be used to measure daily use of the affected upper limb in daily life in this project.The total score ranges from 0 to 30.
Time Frame: Change from baseline at 5 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Robotic Group | Robotic Mirror Group
Number analyzed (Participants) | 14 | 15
score on a scale | 0.15 [0.03 to 0.35] | 0.21 [0.13 to 0.53]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Robotic Group | Robotic Mirror Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT04826900/Prot_SAP_000.pdf